CLINICAL TRIAL: NCT03745820
Title: A Phase 2, Randomized, Double-Blind, Multiple-Dose, Placebo-Controlled Study to Evaluate the Safety and Efficacy of BIIB104 in Subjects With Cognitive Impairment Associated With Schizophrenia (CIAS)
Brief Title: A Study to Evaluate the Safety and Efficacy of BIIB104 in Participants With Cognitive Impairment Associated With Schizophrenia (CIAS)
Acronym: TALLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 263CS201; 2018-003825-27 (EudraCT Number)
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Impairment Associated With Schizophrenia
MeSH Terms: interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIIB104 0.5 mg (Experimental): Participants will receive 0.5 mg of BIIB104 twice a day, orally, for 12 weeks.
  Interventions: Drug: BIIB104
- BIIB104 0.15 mg (Experimental): Participants will receive 0.15 mg of BIIB104 twice a day, orally, for 12 weeks.
  Interventions: Drug: BIIB104
- Matching Placebo (Placebo Comparator): Participants will receive matching placebo twice a day, orally, for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BIIB104 — Administered as specified in the treatment arm
  Other Names: PF-04958242
  Arms: BIIB104 0.15 mg; BIIB104 0.5 mg
Other: Placebo — Administered as specified in the treatment arm
  Arms: Matching Placebo

SUMMARY:
The primary objective of the study is to evaluate the efficacy of BIIB104 in participants with CIAS, using the Working Memory Domain of the MATRICS Consensus Cognitive Battery (MCCB).

The secondary objectives of this study are to evaluate the safety and tolerability of BIIB104 in participants with CIAS, and to evaluate the efficacy of BIIB104 in participants with CIAS on measures of cognition, functioning, and psychiatric symptomology.

ELIGIBILITY:
Key Inclusion Criteria:

* Otherwise healthy participant with a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), diagnosis of schizophrenia of at least 2 years' duration as confirmed by the mini-international neuropsychiatric interview (MINI) 7.0.2 for Psychotic Disorders.
* Evidence of stable schizophrenia symptomatology ≥12 weeks (e.g., no hospitalizations for schizophrenia, no increase in level of psychiatric care due to worsening of schizophrenia symptoms).
* Participants must be in ongoing maintenance atypical antipsychotic therapy (except clozapine), on a stable treatment regimen for ≥8 weeks prior to Baseline/Day 1, including concomitant psychotropic medication. Doses of background atypical antipsychotics should be within the recommended dose range listed in the approved product labeling of the country where the study is being conducted.
* SCI-PANSS: No more than moderate-severe rating (score ≤5) on delusions, hallucinatory behavior, grandiosity, suspiciousness / persecution, and hostility (i.e. PANSS, positive symptom items P1, P3, P5, P6, P7); or unusual thought content (G9); and no more than a moderate rating (score ≤4) on conceptual disorganization (P2).

Key Exclusion Criteria:

* Participation in a trial using any component or version of the MATRICS Consensus Cognitive Battery (MCCB) or the University of California, San Diego (UCSD) Performance-Based Skills Assessment test within the previous 6 months.
* Participation in cognitive remediation therapy within 6 months prior to randomization.
* Screening MCCB Working Memory Domain T-score ≥60.
* Current DSM-5 diagnosis of schizoaffective disorder on the MINI 7.0.2 for Psychotic Disorders.
* Current DSM-5 diagnosis of major depressive episode, manic and hypomanic episode, panic disorder, agoraphobia, social anxiety disorder, obsessive-compulsive disorder, posttraumatic stress disorder, and/or generalized anxiety disorder on the MINI 7.0.2 for Psychotic Disorders.
* Lifetime DSM-5 diagnosis of antisocial personality disorder, anorexia nervosa, bulimia nervosa, and/or binge-eating disorder on the MINI 7.0.2 for Psychotic Disorders.
* Meets the DSM-5 diagnosis of moderate or severe substance use disorder (excluding nicotine dependence) within 12 months of screening on the MINI 7.0.2 for Psychotic Disorders interview.
* DSM-5 diagnosis of Intellectual Disability (intellectual developmental disorder).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (60):
- United States (37):
  - Pillar Clinical Research, LLC, Bentonville, Arkansas
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - Research Site, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - Excell Research, Oceanside, California
  - Research Site, Pico Rivera, California
  - CNRI - San Diego, LLC, San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Research Site, San Diego, California
  - Research Site, San Rafael, California
  - Research Site, Torrance, California
  - Yale University, Department of Psychiatry, New Haven, Connecticut
  - Research Site, Lauderhill, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Chicago, Illinois
  - Alexian Brothers Hospital Network, Hoffman Estates, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - Research Site, Gaithersburg, Maryland
  - Cherry Health, Grand Rapids, Michigan
  - Research Site, Flowood, Mississippi
  - Research Site, St Louis, Missouri
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - UB Department Psychiatry, Buffalo, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - The Ohio State University Department of Psychiatry, Columbus, Ohio
  - Research Site, North Canton, Ohio
  - Research Site, Richardson, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Research Site, Kirkland, Washington
- Germany (4):
  - Zentrum für klinische Forschung Dr. med. I. Schöll, Bad Homburg, Hesse
  - Clinic for Psychiatrie, Frankfurt am Main, Hesse
  - Universitätsmedizin Göttingen, Klinik für Psychiatrie und Psychotherapie, Westerstede, Lower Saxony
  - Dpt of Psychiatry and Psychotherapy, University of Leipzig, Leipzig, Saxony
- Japan (9):
  - Research Site, Anan-shi
  - Research Site, Ichikawa-shi
  - Research Site, Kashihara-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kita-gun
  - Research Site, Kodaira-shi
  - Research Site, Kumagaya-shi
  - Research Site, Takasaki-shi
  - Research Site, Yokosuka-shi
- Spain (7):
  - Hospital Universitario Marques Valdecilla, Santander, Cantabria
  - Research Site, Majadahonda, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Unidad Neurociencias CS San Juan, Salamanca
  - Research Site, Seville
- United Kingdom (3):
  - Oxford Health NHS Foundation Trust, Oxford, Oxfordshire
  - Abraham Cowley Unit, Lyne, Surrey
  - Research Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 53 investigative sites in the United States, Japan, Spain, Germany, and the United Kingdom from 15 Nov 2018 to 07 April 2022.
Pre-assignment Details: A total of 554 participants were screened out of which, 195 participants were randomized and dosed to receive BIIB104 or placebo.
Groups:
- Placebo: Participants received BIIB104 matching placebo capsules, twice a day (BID), orally for 12 weeks.
- BIIB104 0.15 mg: Participants received 0.15 milligrams (mg) capsules of BIIB104, BID, orally for 12 weeks.
- BIIB104 0.5 mg: Participants received 0.5 mg capsules of BIIB104, BID, orally for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Started | 64 | 66 | 65
Safety Analysis Set (The safety population included all randomized participants who received at least 1 dose of study treatment(BIIB104 or placebo). One participant randomized to placebo, inadvertently received one or more doses of active treatment.) | 63 | 66 | 66
Completed | 52 | 52 | 51
Not Completed | 12 | 14 | 14
Not completed — Adverse Event | 0 | 3 | 2
Not completed — Non-Compliance with Study Drug | 4 | 3 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 4
Not completed — Physician decision unrelated to safety/efficacy | 0 | 0 | 4
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Reason not Specified | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least one dose of study treatment (BIIB104 or placebo).
Groups:
- Placebo: Participants received BIIB104 matching placebo capsules, BID, orally for 12 weeks.
- BIIB104 0.15 mg: Participants received 0.15 mg capsules of BIIB104, BID, orally for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg | Total
Number analyzed (Participants) | 64 | 66 | 65 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (9.47) | 37.7 (9.41) | 41.3 (9.63) | 39.8 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 18 | 59
  Male | 44 | 45 | 47 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 6 | 25
  Not Hispanic or Latino | 45 | 47 | 49 | 141
  Unknown or Not Reported | 9 | 10 | 10 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10 | 8 | 13 | 31
  Black or African American | 29 | 27 | 26 | 82
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  White | 15 | 19 | 15 | 49
  Other | 0 | 2 | 0 | 2
  Unknown | 9 | 10 | 10 | 29
MATRICS Consensus Cognitive Battery (MCCB) Working Memory Domain Score [Mean (Full Range); unit: score on a scale] — The MCCB is a cognitive battery that assesses 7 domains recommended by the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) initiative (i.e., Working Memory, Verbal Learning, Speed of Processing, Attention/Vigilance, Visual Learning, Social Cognition, and Reasoning and Problem Solving). MCCB was administered via laptop computer and paper-and-pencil assessments. MCCB composite T scores are between 40 and 60 (normal range). Higher scores indicate better cognitive functioning. The working memory domain score of the MCCB is reported.
  score on a scale | 39.6 [17 to 70] | 38.5 [12 to 60] | 39.8 [17 to 58] | 39.3 [12 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Change From Baseline in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Working Memory Domain Score at Week 12
Description: The MCCB is a cognitive battery that assesses 7 domains recommended by the MATRICS initiative (i.e., Working Memory, Verbal Learning, Speed of Processing, Attention/Vigilance, Visual Learning, Social Cognition, and Reasoning and Problem Solving). MCCB was administered via laptop computer and paper-and-pencil assessments. T-scores for the individual tests were calculated according to the developer's recommended scoring algorithms. MCCB composite T scores are between 40 and 60 (normal range). Higher scores indicate better cognitive functioning. The working memory domain score of the MCCB is reported in this outcome measure.
Time Frame: Baseline and Week 12
Population: ITT population included all randomized participants who received at least one dose of study treatment (BIIB104 or placebo). Here, "Overall Number of Participants Analyzed" signifies the number of participants analyzed in this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 50 | 50 | 49
score on a scale | 1.17 (0.939) | 0.91 (0.936) | 0.84 (0.934)
Statistical Analysis 1: Comparison: Placebo vs BIIB104 0.15 mg; Mixed Model Repeated Measures(MMRM)model was used to analyze change from baseline of outcome measure(OM)using fixed effects of treatment group,region,study visit,study visit-by-treatment interaction,baseline value of OM,baseline-by-visit interaction; Test type: Superiority; p = 0.8472, MMRM; Least Squares (LS) Mean Difference = -0.26, 95% CI 2-sided [-2.88 to 2.37], Standard Error of Mean 1.328
Statistical Analysis 2: Comparison: Placebo vs BIIB104 0.5 mg; A MMRM model was used to analyze the change from baseline of the OM of interest, using fixed effects of treatment group, region, study visit, study visit-by-treatment interaction, baseline value of OM, baseline-by-visit interaction; Test type: Superiority; p = 0.8053, MMRM; LS Mean Difference = -0.33, 95% CI 2-sided [-2.94 to 2.29], Standard Error of Mean 1.323

2. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect, or is a medically important event.
Time Frame: From first dose of study drug through end of the study (up to Week 14)
Population: The safety population included all randomized participants who received at least 1 dose of study treatment (BIIB104 or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 63 | 66 | 66
Participants
  AEs | 28 | 32 | 28
  SAEs | 1 | 1 | 2

3. Secondary Outcome: Mean Total Score Assessed by Scale for the Assessment and Rating of Ataxia (SARA)
Description: The SARA is a clinical scale that is based on a semiquantitative assessment of cerebellar ataxia on an impairment level and complements the brief neurological examination. The SARA scale is an eight-item clinical rating scale (gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements, and heel-shin test) with a total score range of 0-40, where 0 is the best neurological status and 40 is the worst neurological status.
Time Frame: Baseline, Weeks 2, 6, 12 and safety follow-up (Week 14)
Population: The safety population included all randomized participants who received at least 1 dose of study treatment (BIIB104 or placebo). Here, "Overall number of participants analyzed" signifies the number of participants analyzed in this outcome measure and "number analyzed" signifies the number of participants analyzed at specified time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 62 | 64 | 65
score on a scale
  Baseline | 0.5 (1.03) | 0.4 (1.15) | 0.3 (0.92)
  Week 2: number analyzed (Participants) | 57 | 59 | 62
  Week 2 | 0.4 (0.85) | 0.5 (1.10) | 0.3 (0.68)
  Week 6: number analyzed (Participants) | 52 | 56 | 60
  Week 6 | 0.4 (0.71) | 0.3 (0.90) | 0.2 (0.58)
  Week 12: number analyzed (Participants) | 52 | 51 | 54
  Week 12 | 0.4 (0.80) | 0.3 (0.82) | 0.2 (0.72)
  Week 14: number analyzed (Participants) | 55 | 58 | 57
  Week 14 | 0.4 (0.85) | 0.3 (0.91) | 0.2 (0.69)

4. Secondary Outcome: Number of Participants With at Least One Event of Suicidal Ideation and/or Suicidal Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. Suicidal ideation is classified on a 5-item scale: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active suicidal ideation with some intent to act, without specific plan), and 5 (active suicidal ideation with specific plan and intent). Suicidal behavior is classified on a 6-item scale: 1 (actual attempt), 2 (interrupted attempt), 3 (aborted attempt), 4 (preparatory acts or behavior), 5 (suicidal behavior), and 6 (suicide). The data analyzed signifies the participants with at least one event of suicidal ideation and/or suicidal behavior.
Time Frame: Up to Week 14
Population: The safety population included all randomized participants who received at least 1 dose of study treatment (BIIB104 or placebo). Here, "Overall Number of Participants Analyzed" signifies the number of participants analyzed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 63 | 65 | 65
Participants | 3 | 4 | 0

5. Secondary Outcome: Change From Baseline in University of California, San Diego Performance Based Skills Assessment-Brief International Version (UPSA-Bi) Assessment at Week 12
Description: The UPSA-Bi, international version, an abbreviated version of the UPSA-Validation of Intermediate Measures, is a measure of functional capacity and assesses skills used in community tasks. This assessment measures 2 general skills that were previously identified as essential to functioning in the community: financial skills and communication skills. The UPSA-Bi assessment is scored from 0-100, higher scores indicating higher functional status.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 49 | 50 | 49
score on a scale | 2.07 (1.303) | 5.50 (1.292) | 5.49 (1.305)
Statistical Analysis 1: Comparison: Placebo vs BIIB104 0.15 mg; An analysis of covariance (ANCOVA) model was applied adjusting for treatment group and baseline value of the OM; Test type: Superiority; p = 0.0637, ANCOVA; LS Mean Difference = 3.43, 95% CI 2-sided [-0.20 to 7.06], Standard Error of Mean 1.835
Statistical Analysis 2: Comparison: Placebo vs BIIB104 0.5 mg; An ANCOVA model was applied adjusting for treatment group and baseline value of the OM; Test type: Superiority; p = 0.0659, ANCOVA; LS Mean Difference = 3.42, 95% CI 2-sided [-0.23 to 7.06], Standard Error of Mean 1.844

6. Secondary Outcome: Change From Baseline in Schizophrenia Cognition Rating Scale (SCoRS) Assessment Score at Week 12
Description: The SCoRS is an interview-based assessment of cognition that involves interviews with participants and informants. The SCoRS includes 20 items designed to specifically assess aspects of cognitive functioning found in each of the seven MCCB cognitive domains including the following: Memory: 4 items; Learning: 2 items; Attention: 3 items; Working memory: 2 items; Problem solving: 3 items; Processing/motor speed: 2 items; Social cognition: 3 items; Language: 1 item. Total score range is 20-80, lower scores indicating higher functional status. The data reported in this outcome measure are for global rating score.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 49 | 48 | 50
score on a scale | -0.51 (0.146) | -0.42 (0.148) | -0.41 (0.145)
Statistical Analysis 1: Comparison: Placebo vs BIIB104 0.15 mg; An ANCOVA model was applied adjusting for treatment group and baseline value of the OM; Test type: Superiority; p = 0.6653, ANCOVA; LS Mean Difference = 0.208, 95% CI 2-sided [-0.32 to 0.50], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs BIIB104 0.5 mg; An ANCOVA model was applied adjusting for treatment group and baseline value of the OM; Test type: Superiority; p = 0.6140, ANCOVA; LS Mean Difference = 0.206, 95% CI 2-sided [-0.30 to 0.51], Standard Error of Mean 0.10

7. Secondary Outcome: Change From Baseline in MCCB Neurocognitive Composite Scores at Week 12
Description: The MCCB is a cognitive battery that assesses 7 domains recommended by the MATRICS initiative (i.e., Working Memory, Verbal Learning, Speed of Processing, Attention/Vigilance, Visual Learning, Social Cognition, and Reasoning and Problem Solving). MCCB was administered via laptop computer and paper-and-pencil assessments. T-scores for the individual tests were calculated according to the developer's recommended scoring algorithms. MCCB composite T scores are between 40 and 60 (normal range). Higher scores indicate better cognitive functioning. The MCCB composite score contains all of the tests and domains of the MCCB.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 50 | 50 | 49
score on a scale | 2.90 (0.733) | 1.80 (0.728) | 3.39 (0.727)
Statistical Analysis 1: Comparison: Placebo vs BIIB104 0.15 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.2886, MMRM; LS Mean Difference = -1.10, 95% CI 2-sided [-3.14 to 0.94], Standard Error of Mean 1.033
Statistical Analysis 2: Comparison: Placebo vs BIIB104 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.6349, MMRM; LS Mean Difference = 0.49, 95% CI 2-sided [-1.55 to 2.53], Standard Error of Mean 1.032

8. Secondary Outcome: Change From Baseline in MCCB Individual Domain Scores (Excluding Working Memory Domain) at Week 12
Description: The MCCB is a cognitive battery that assesses 7 domains recommended by the MATRICS initiative (i.e., working memory, verbal learning, speed of processing, attention/vigilance, visual learning, social cognition, and reasoning and problem solving). MCCB was administered via laptop computer and paper-and-pencil assessments. T-scores for the individual tests were calculated according to the developer's recommended scoring algorithms. MCCB composite T scores are between 40 and 60 (normal range). Higher scores indicate better cognitive functioning. All the domain scores of the MCCB are reported in this outcome measure with the exception of working memory domain.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 50 | 50 | 49
score on a scale
  Verbal Learning: Change at Week 12 | 0.95 (0.951) | 1.41 (0.946) | 0.41 (0.950)
  Speed of Processing: Change at Week 12 | 4.42 (0.824) | 2.28 (0.819) | 3.99 (0.817)
  Attention/Vigilance: Change at Week 12 | 0.62 (0.852) | 0.53 (0.848) | 1.55 (0.848)
  Visual Learning: Change at Week 12 | 1.70 (1.131) | 0.19 (1.125) | 1.77 (1.125)
  Social Cognition: Change at Week 12 | -0.13 (0.959) | 1.06 (0.953) | 0.95 (0.955)
  Reasoning and Problem Solving: Change at Week 12 | 2.81 (1.019) | 2.10 (1.1014) | 4.40 (1.011)
Statistical Analysis 1: Comparison: Placebo vs BIIB104 0.15 mg; Verbal Learning: Change From Baseline at Week 12; Test type: Superiority; p = 0.7372, MMRM — A MMRM model was used to analyze the change from baseline of the OM of interest, using fixed effects of treatment group, region, study visit, study visit-by-treatment interaction, baseline value of OM, baseline-by-visit interaction; LS Mean Difference = 0.45, 95% CI 2-sided [-2.21 to 3.11], Standard Error of Mean 1.345
Statistical Analysis 2: Comparison: Placebo vs BIIB104 0.5 mg; Verbal Learning: Change From Baseline at Week 12; Test type: Superiority; p = 0.6894, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.54, 95% CI 2-sided [-3.20 to 2.12], Standard Error of Mean 1.346
Statistical Analysis 3: Comparison: Placebo vs BIIB104 0.15 mg; Speed of Processing: Change From Baseline at Week 12; Test type: Superiority; p = 0.0674, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -2.14, 95% CI 2-sided [-4.44 to 0.16], Standard Error of Mean 1.162
Statistical Analysis 4: Comparison: Placebo vs BIIB104 0.5 mg; Speed of Processing: Change From Baseline at Week 12; Test type: Superiority; p = 0.7132, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.43, 95% CI 2-sided [-2.72 to 1.87], Standard Error of Mean 1.161
Statistical Analysis 5: Comparison: Placebo vs BIIB104 0.15 mg; Attention/Vigilance: Change From Baseline at Week 12; Test type: Superiority; p = 0.9428, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.09, 95% CI 2-sided [-2.46 to 2.29], Standard Error of Mean 1.203
Statistical Analysis 6: Comparison: Placebo vs BIIB104 0.5 mg; Attention/Vigilance: Change From Baseline at Week 12; Test type: Superiority; p = 0.4425, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.93, 95% CI 2-sided [-1.45 to 3.30], Standard Error of Mean 1.202
Statistical Analysis 7: Comparison: Placebo vs BIIB104 0.15 mg; Visual Learning: Change From Baseline at Week 12; Test type: Superiority; p = 0.3455, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.51, 95% CI 2-sided [-4.66 to 1.64], Standard Error of Mean 1.597
Statistical Analysis 8: Comparison: Placebo vs BIIB104 0.5 mg; Visual Learning: Change From Baseline at Week 12; Test type: Superiority; p = 0.9686, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 0.06, 95% CI 2-sided [-3.09 to 3.21], Standard Error of Mean 1.595
Statistical Analysis 9: Comparison: Placebo vs BIIB104 0.15 mg; Social Cognition: Change From Baseline at Week 12; Test type: Superiority; p = 0.3832, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 1.18, 95% CI 2-sided [-1.49 to 3.85], Standard Error of Mean 1.351
Statistical Analysis 10: Comparison: Placebo vs BIIB104 0.5 mg; Social Cognition: Change From Baseline at Week 12; Test type: Superiority; p = 0.4297, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean DIfference = 1.07, 95% CI 2-sided [-1.61 to 3.75], Standard Error of Mean 1.357
Statistical Analysis 11: Comparison: Placebo vs BIIB104 0.15 mg; Reasoning and Problem Solving: Change From Baseline at Week 12; Test type: Superiority; p = 0.6245, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.71, 95% CI 2-sided [-3.55 to 2.14], Standard Error of Mean 1.438
Statistical Analysis 12: Comparison: Placebo vs BIIB104 0.5 mg; Reasoning and Problem Solving: Change From Baseline at Week 12; Test type: Superiority; p = 0.2698, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = 1.59, 95% CI 2-sided [-1.25 to 4.43], Standard Error of Mean 1.436

9. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score, Positive Subscale, and Negative Subscale Scores at Week 12
Description: The PANSS includes 3 subscales and 30 items: 7 items that make up the Positive subscale (e.g., delusions, conceptual disorganization, hallucinatory behaviour); 7 items that make up the Negative subscale (e.g., blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal); and 16 items that make up the General Psychopathology subscale (e.g., somatic concern, anxiety, guilt feelings, mannerisms and posturing, motor retardation, uncooperativeness, disorientation, poor impulse control, preoccupation). Each item on the positive, negative and general psychopathology subscale is rated from 1 (absent) to 7 (extreme). The score range is 7-49 for positive and negative subscales, score range is 16-112 for the general psychopathology subscale. Total PANSS score (positive+ negative + general psychopathology subscale scores) range from 30 to 210. Higher scores represent more severity in symptoms.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 51 | 51 | 50
score on a scale
  Positive Symptoms Subscale: Change From Baseline at Week 12 | -0.65 (0.431) | -1.09 (0.430) | -0.98 (0.429)
  Negative Symptoms Subscale: Change From Baseline at Week 12 | -0.90 (0.461) | -0.98 (0.461) | -1.40 (0.460)
  Total Score: Change From Baseline at Week 12 | -3.06 (1.429) | -4.26 (1.421) | -5.03 (1.427)
Statistical Analysis 1: Comparison: Placebo vs BIIB104 0.15 mg; Positive Symptoms Subscale: Change From Baseline at Week 12; Test type: Superiority; p = 0.4654, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.45, 95% CI 2-sided [-1.65 to 0.76], Standard Error of Mean 0.610
Statistical Analysis 2: Comparison: Placebo vs BIIB104 0.5 mg; Positive Symptoms Subscale: Change From Baseline at Week 12; Test type: Superiority; p = 0.5886, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.33, 95% CI 2-sided [-1.53 to 0.87], Standard Error of Mean 0.608
Statistical Analysis 3: Comparison: Placebo vs BIIB104 0.15 mg; Negative Symptoms Subscale: Change From Baseline at Week 12; Test type: Superiority; p = 0.9079, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.08, 95% CI 2-sided [-1.37 to 1.22], Standard Error of Mean 0.655
Statistical Analysis 4: Comparison: Placebo vs BIIB104 0.5 mg; Negative Symptoms Subscale: Change From Baseline at Week 12; Test type: Superiority; p = 0.4441, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -0.50, 95% CI 2-sided [-1.78 to 0.79], Standard Error of Mean 0.650
Statistical Analysis 5: Comparison: Placebo vs BIIB104 0.15 mg; Total Score: Change From Baseline at Week 12; Test type: Superiority; p = 0.5537, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.20, 95% CI 2-sided [-5.18 to 2.79], Standard Error of Mean 2.017
Statistical Analysis 6: Comparison: Placebo vs BIIB104 0.5 mg; Total Score: Change From Baseline at Week 12; Test type: Superiority; p = 0.3320, MMRM — [p-value comment as in outcome 8, analysis 1]; LS Mean Difference = -1.96, 95% CI 2-sided [-5.95 to 2.02], Standard Error of Mean 2.018

10. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scores at Week 12
Description: The CGI-S consists of a single 7-point rating score of illness severity. The following question: "Considering your total clinical experience with this particular population, how mentally ill is your participant at this time?" is rated with a score from 1 to 7- 1: Normal, not ill at all; 2: Borderline mentally ill; 3: Mildly ill; 4: Moderately ill; 5: Markedly ill; 6: Severely ill; or 7: Among the most severely ill participants. Lower scores indicate less severity of illness.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 51 | 50 | 50
score on a scale | -0.19 (0.091) | -0.16 (0.091) | -0.19 (0.091)
Statistical Analysis 1: Comparison: Placebo vs BIIB104 0.15 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.8517, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.23 to 0.28], Standard Error of Mean 0.128
Statistical Analysis 2: Comparison: Placebo vs BIIB104 0.5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.9952, MMRM; LS Mean Difference = 0.00, 95% CI 2-sided [-0.25 to 0.25], Standard Error of Mean 0.128

11. Secondary Outcome: Number of Participants With Response on Clinical Global Impression-Improvement (CGI-I) Scale at Week 12
Description: The CGI-I consists of a single 7-point rating score total improvement, regardless of whether or not the change is due entirely to drug treatment. The following question: "Compared to your participant's condition at the beginning of treatment, how much has your participant changed?" is rated with a score from 1 to 7- 1: Very much improved; 2: Much improved; 3: Minimally improved; 4: No change; 5: Minimally worse; 6: Much worse; or 7: Very much worse. Lower scores indicate greater improvement.
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
Number analyzed (Participants) | 51 | 50 | 50
Participants
  Very Much Improved | 1 | 1 | 0
  Much Improved | 11 | 4 | 4
  Minimally Improved | 13 | 18 | 18
  No Change | 22 | 26 | 26
  Minimally Worse | 2 | 1 | 2
  Much Worse | 2 | 0 | 0
  Very Much Worse | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of the study (up to Week 14)
Description: The safety population included all randomized participants who received at least 1 dose of study treatment(BIIB104 or placebo).One participant randomized to placebo,inadvertently received one or more doses of active treatment. For participants affected, a participant was counted only once within each system organ class/preferred term/study period.
Arm/Group | Placebo | BIIB104 0.15 mg | BIIB104 0.5 mg
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/63 | 1/66 | 2/66
Other Adverse Events (participants affected / at risk) | 2/63 | 2/66 | 8/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=63) | BIIB104 0.15 mg (N=66) | BIIB104 0.5 mg (N=66)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
Psychiatric decompensation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=63) | BIIB104 0.15 mg (N=66) | BIIB104 0.5 mg (N=66)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Schizophrenia (Psychiatric disorders) | 1 (1) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03745820/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03745820/SAP_001.pdf